CLINICAL TRIAL: NCT04078555
Title: A Randomized, Double-Blind, Placebo-controlled, Parallel, Phase II Study to Evaluate Efficacy and Safety of ENERGI-F703 GEL in Subjects With Venous Leg Ulcer (VLU)
Brief Title: A Study to Evaluate ENERGI-F703 GEL in Venous Leg Ulcer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Energenesis Biomedical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ENERGI-F703-02
Record Dates: First submitted 2019-08-28; First posted 2019-09-06 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Venous Leg Ulcer
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ENERGI-F703 GEL (Experimental): topical application on target venous leg ulcer, twice daily
  Interventions: Drug: ENERGI-F703 GEL
- ENERGI-F703 GEL matched vehicle (Placebo Comparator): topical application on target venous leg ulcer, twice daily
  Interventions: Drug: ENERGI-F703 GEL matched vehicle

INTERVENTIONS:
Drug: ENERGI-F703 GEL — The study medication will be applied twice daily until the end of 84 days or up to the visit confirmation of complete ulcer closure, whichever comes first.
  The estimated amount of study medication applied to the ulcer area is 0.25 cm (about 0.11 g) in length per cm2 of ulcer size.
  Arms: ENERGI-F703 GEL
Drug: ENERGI-F703 GEL matched vehicle — The study medication will be applied twice daily until the end of 84 days or up to the visit confirmation of complete ulcer closure, whichever comes first.
  The estimated amount of study medication applied to the ulcer area is 0.25 cm (about 0.11 g) in length per cm2 of ulcer size.
  Arms: ENERGI-F703 GEL matched vehicle

SUMMARY:
This is a randomized, double-blind, placebo-controlled, phase II, multi-centered study to evaluate the efficacy and safety of ENERGI-F703 GEL in subjects who are ≥ 20 years old with venous leg ulcer (VLU). Subjects will be recruited from multiple sites in Taiwan. The treatment period will be 84 days with another 84-day follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. With either gender aged at least 20 years old
2. With venous reflux >0.1 sec measured by duplex ultrasound imaging dated within 6 months prior to the Screening visit
3. With at least one venous ulcer on the lower leg (knee to ankle inclusive) and not healing for at least 4 weeks. The ulcer with the largest surface area will be selected as target ulcer. If two or more ulcers have the largest size, the one with the longest duration will be selected
4. With the target ulcer size of 2 cm2 to 50 cm2
5. Target VLU involves a full thickness skin loss, but without exposure of tendon, muscle, or bone
6. Target VLU should be free of any necrosis or infection in any soft tissue and bone tissue
7. Able to tolerate compression therapy
8. Subject has signed the written informed consent form

Exclusion Criteria:

1. Target VLU With active cellulitis or osteomyelitis
2. With target ulcer size decreased by at least 30% after 2 weeks of standard care
3. With poor nutritional status (albumin < 2g/dl), poor diabetic control (HbA1c > 12%), a leukocyte counts < 2,000/mm3, abnormal liver function (AST, ALT>3 × upper limit of normal range) tests within 14 days prior to Screening visit or 28 days prior to Randomization visit
4. Requiring treatment with chemotherapeutic agents
5. With known or suspected hypersensitivity to any ingredients of IP and matched vehicle
6. With coronary heart disease with myocardial infarction, coronary artery bypass graft (CABG), or percutaneous transluminal coronary angioplasty (PTCA) within 3 months prior to Screening visit
7. (1) Female subject of childbearing potential who:

   * is lactating; or
   * has positive pregnancy test result at eligibility checking; or
   * refuses to adopt at least one form of birth control from signing informed consent to the end of study

   Note:

   Acceptable forms include:

   Established use of oral, injected or implanted hormonal methods of contraception. Placement of an intrauterine device (IUD) or intrauterine system (IUS).Barrier methods of contraception: Condom OR Occlusive cap (diaphragm or cervical/vault caps)

   7(2) Male subject with female spouse/partners who are of childbearing potential refuses to adopt at least one form of birth control (at least one of which must be a barrier method) from signing informed consent to the end of study)
8. With ankle brachial index (ABI) < 0.6
9. Enrollment in any investigational drug trial within 4 weeks before entering this study
10. With any condition judged by the investigator that entering the trial may be detrimental to the subject

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-07-26 (Actual); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of complete ulcer closure | Day -21 to Day 99
  Complete wound closure is defined as 100% skin re-epithelialization without drainage or dressing requirements confirmed at two consecutive study visit 2 weeks apart.

SECONDARY OUTCOMES:
Percentage change in target ulcer area from baseline to each post-treatment visit | Day -21 to Day 85
Time-to-Complete ulcer closure of target ulcer | Day -21 to Day 99
  Complete wound closure is defined as 100% skin re-epithelialization without drainage or dressing requirements confirmed at two consecutive study visit 2 weeks apart.
The accumulated confirmed target ulcer closure incidence at each of the post-treatment visit | Day -21 to Day 85
  Complete wound closure is defined as 100% skin re-epithelialization without drainage or dressing requirements confirmed at two consecutive study visit 2 weeks apart.
Incidence of vital signs abnormalities | Day -21 to Day 169
  Vital signs measurement will consist of systolic/diastolic blood pressure, respiratory rate, pulse rate or heart rate, and body temperature.
Incidence of physical examination abnormalities | Day -21 to Day 169
  Physical examination will include the following items: general appearance, skin, eyes, ears, nose, throat, head and neck, heart, chest and lungs, abdomen, extremities, lymph nodes, musculoskeletal, neurological and others.
Incidence of laboratory examination results abnormalities | Day -21 to Day 169
  The laboratory examinations include Hematology tests (CBC), Biochemistry (AST, ALP, ALT, serum creatinine, BUN, albumin and fasting glucose) and Urinalysis (pH, glucose, RBC, WBC and protein).
Incidence of AEs and SAEs | Day -21 to Day 169

CONTACTS AND LOCATIONS:
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan